CLINICAL TRIAL: NCT05504746
Title: A Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of SHEN26 Capsule in Healthy Participants
Brief Title: A Phase I Study of SHEN26 Capsule in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Kexing Pharmaceutical Co., Ltd. (Network)
Responsible Party: Sponsor
Organization: Kexing Biopharm Co., Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KXZY-SHEN26-101
Record Dates: First submitted 2022-08-10; First posted 2022-08-17 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SHEN26 capsule (SAD and FE part) (Experimental): SHEN26 capsule 50mg, 200mg, 400mg, 800mg, and 1200mg dose groups
  Interventions: Drug: SHEN26 capsule
- SHEN26 capsule (MAD part) (Experimental): SHEN26 capsule 200mg, 400mg, and 600mg dose groups
  Interventions: Drug: SHEN26 capsule
- SHEN26 placebo (SAD and FE part) (Placebo Comparator): SHEN26 placebo 50mg, 200mg, 400mg, 800mg, and 1200mg dose groups
  Interventions: Drug: SHEN26 placebo
- SHEN26 placebo (MAD part) (Placebo Comparator): SHEN26 placebo 200mg, 400mg, and 600mg dose groups
  Interventions: Drug: SHEN26 placebo

INTERVENTIONS:
Drug: SHEN26 capsule — Specification: 50mg/capsule and 200mg/capsule. Participants will receive SHEN26 capsule(s) orally for a single dose.
  The specification of 50mg/capsule will only be used for the 50mg dose group in the SAD part. For the other dose groups and other parts of the study, 200mg/capsule will be used.
  Arms: SHEN26 capsule (SAD and FE part)
Drug: SHEN26 capsule — Specification: 200mg/capsule. Participants will receive SHEN26 capsules orally for Q12h X 5.5 days.
  Arms: SHEN26 capsule (MAD part)
Drug: SHEN26 placebo — Placebo matching the SHEN26 capsule. Specification: 50mg/capsule and 200mg/capsule.
  Participants will receive SHEN26 placebo orally for a single dose.
  Arms: SHEN26 placebo (SAD and FE part)
Drug: SHEN26 placebo — Placebo matching the SHEN26 capsule. Specification: 200mg/capsule.
  Participants will receive SHEN26 placebo orally for Q12h X 5.5 days.
  Arms: SHEN26 placebo (MAD part)

SUMMARY:
This is a randomized, double-blind, and placebo-controlled phase I clinical trial. It is designed to assess the safety, tolerability, and pharmacokinetic (PK) profile of SHEN26 capsules after single and multiple ascending dosing in healthy Chinese adult participants, and the food effect on the PK profile of SHEN26 capsules.

DETAILED DESCRIPTION:
This phase of the study includes three parts: single ascending dose (SAD), food effect (FE), and multiple ascending dose (MAD) in healthy participants.

* SAD Part: There are dose groups of 50 mg, 200 mg, 400 mg, 800 mg, and 1200 mg for the SAD part of the trial.
* FE Part: This part of the study is tentatively assigned to the 400 mg dose group of the SAD part. After the participants complete the SAD part and pass their safety check on Day 4, they enter the second cycle. Participants are required to fast for more than 10 hours on the night of Day 4, and they will be dosed again on Day 5, 30 min after the start of the high-fat meal (the meal had to be completed within 30 min).
* MAD Part: Based on the safety, tolerability, and PK data from the SAD part, if available, the appropriate dose will be selected for the MAD study. Three dose groups of 200 mg, 400 mg, and 600 mg are planned for this part of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants aged 18-45 years (including boundary values, based on the time of signing the informed consent);
2. Body mass index (BMI) within the range of 19.0-26.0 kg/m^2 (including boundary values), with body weight of not less than 50.0 kg for males and 45.0 kg for females;
3. Participants were evaluated by the investigator on the basis of their medical history, physical examination, vital signs, 12-lead electrocardiogram, laboratory tests (CBC, CMP, urinalysis, urine microalbumin test, urinary NAG test, coagulation test, serum virology, blood alcohol content, drug abuse screening test, and blood pregnancy test, etc.), abdominal ultrasound, ophthalmologic examination, and chest CT for overall good health status (normal or abnormal test results without clinical significance);
4. Fully understand the purpose, nature, methods, and possible adverse events of the trial, volunteer as a participant, and sign an informed consent form;
5. The participant and their female partner have no birth plan and voluntarily use effective contraception methods and have no plans to donate sperm or eggs from 2 weeks prior to screening until 6 months after the last dose of the study drug, and to ensure the use of one or more non-pharmacological contraceptive methods during sexual intercourse from 2 weeks prior to screening until 1 month after the last dose of the study drug.

Exclusion Criteria:

1. Persons with pre-screening or ongoing disease with abnormal clinical manifestations to be excluded, including but not limited to diseases of the nervous/psychiatric system, respiratory system, cardiovascular system, digestive system (any history of gastrointestinal disorders affecting drug absorption), hematologic and lymphatic system, urinary system, endocrine system, and immune system；
2. Persons with a history of febrile illness within 14 days prior to screening；
3. Persons with dysphagia, history of gastrointestinal surgery or other related medical conditions that may interfere with the absorption and/or elimination of oral medications；
4. Persons who have undergone major surgical procedures (excluding diagnostic surgery) within 3 months prior to screening that, in the judgment of the investigator, may interfere with this trial, or who are expected to require major surgery during the trial;
5. Persons who have used or anticipate using any drug that induces or inhibits hepatic metabolic enzymes from 28 days prior to screening through the end of the trial;
6. Persons who have used or expect to use inhibitors of BCRP prior to screening up to 72 h after the last dose;
7. Persons who have used or expect to use inhibitors or inducers of P-gp prior to screening up to 72 h after the last dose;
8. Persons who have used any prescription, over-the-counter, herbal or nutraceutical drug within 14 days prior to screening;
9. Persons who have a history of substance abuse within 5 years prior to screening or who have used drugs in the 3 months prior to screening;
10. Persons with a history of drug or other allergies, particularly to the test drug or any component of the test drug;
11. Persons who have received any vaccine within 1 month prior to screening or who are scheduled to receive a vaccine during the trial;
12. Persons who have a history of blood donation or blood loss of more than 400 mL within 3 months prior to screening, or plan to donate blood during the trial;
13. Persons who have participated in other drug clinical trials and used other clinical trial drugs within 3 months prior to screening;
14. Persons who have difficulties with venous blood collection or have a history of dizziness from needles and blood;
15. Persons who smoked more than 5 cigarettes per day or habitually used nicotine-containing products within 3 months prior to screening, or cannot discontinue use of any tobacco product during the trial;
16. Persons who have consumed more than 14 units of alcohol per week (1 unit of alcohol = 360 mL of beer or 45 mL of 40% alcohol spirits or 150 mL of wine) within 3 months prior to screening or have consumed alcohol-containing products 48 h prior to receiving the test drug, or are unable to abstain from alcohol during the trial;
17. Persons who have ingested any food or beverage containing or metabolized to produce caffeine or xanthine (e.g., coffee, tea, chocolate) within 48 h prior to the administration of the drug;
18. Persons who have taken any food or beverage containing enzymes that induce or inhibit liver metabolism (e.g. grapefruit, etc.) within 7 days prior to recruitment;
19. Persons who have special dietary requirements and cannot accept a unified diet;
20. Female participants who are pregnant or breastfeeding during the trial;
21. Persons who have a positive SARS-CoV-2 test result (oropharyngeal swab PCR test);
22. Any other circumstances that, in the opinion of the investigator, may affect the participant's ability to provide informed consent or follow the trial protocol, or the participant's participation in the trial may affect the trial results or their own safety.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2022-12-11 (Actual)

PRIMARY OUTCOMES:
AEs and SAEs | From Screening period up to Day 12
  The incidence and severity of adverse events (AEs) and serious adverse events (SAEs).
The Number and Percentage of Participants With Clinically Significant Abnormal Vital Signs | From Screening period up to Day 12
  Vital Signs: blood pressure (systolic and diastolic), pulse, body temperature (ear temperature), and respiratory rate. The number and percentage of participants with clinically significant abnormal vital signs will be noted.
The Number and Percentage of Participants With Clinically Significant Abnormal Physical Examination Results | From Screening period up to Day 12
  Physical Examination: skin, lymph nodes, head and neck, chest, abdomen, spine/extremities/joints, and nervous system. The number and percentage of participants with clinically significant abnormal physical examination results will be noted.
The Number and Percentage of Participants With Clinically Significant Abnormal Laboratory Values | From Screening period up to Day 12
  Laboratory Tests: CBC test, CMP test, urinalysis, urine microalbumin test, urinary NAG test, coagulation test, etc. The number and percentage of participants with clinically significant abnormal laboratory values will be noted.
The Number and Percentage of Participants With Clinically Significant Abnormal Abdominal Ultrasound Results | From Screening period up to Day 12
  The number and percentage of participants with clinically significant abnormal abdominal ultrasound imaging test results, including liver, gallbladder, pancreas, spleen, and kidney, will be noted.
The Number and Percentage of Participants With Clinically Significant Abnormal Ophthalmology Examination Results | From Screening period up to Day 12
  Ophthalmology Examination: slit lamp examination. The number and percentage of participants with clinically significant abnormal ophthalmological test results will be noted.
The Number and Percentage of Participants With Clinically Significant Abnormal 12-lead Electrocardiogram (ECG) Values | From Screening period up to Day 12
  12-lead Electrocardiogram (ECG): heart rate, PR, QRS, QT, and QTcF intervals. The number and percentage of participants with clinically significant abnormal 12-lead Electrocardiogram (ECG) values will be noted.

SECONDARY OUTCOMES:
Cmax After a Single Dose of SHEN26 capsule | From predose to 72 hours postdose
  The maximum concentration (Cmax) of SHEN26 capsule.
Tmax After a Single Dose of SHEN26 capsule | From predose to 72 hours postdose
  The time to the maximum concentration (Tmax) of SHEN26 capsule.
AUC0-t and AUC0-inf After a Single Dose of SHEN26 capsule | From predose to 72 hours postdose
  The area under the concentration-time curve (AUC0-t and AUC0-inf) of SHEN26 capsule.
t1/2 After a Single Dose of SHEN26 capsule | From predose to 72 hours postdose
  The elimination half-life (t1/2) of SHEN26 capsule.
CL/F After a Single Dose of SHEN26 capsule | From predose to 72 hours postdose
  The apparent clearance (CL/F) of SHEN26 capsule.
Vz/F After a Single Dose of SHEN26 capsule | From predose to 72 hours postdose
  The apparent volume of distribution (Vz/F) of SHEN26 capsule.
Ke After a Single Dose of SHEN26 capsule | From predose to 72 hours postdose
  The elimination rate constant (Ke) of SHEN26 capsule.
Ae After a Single Dose of SHEN26 capsule | From predose to 72 hours postdose
  (For SAD 400mg dose group only) The amount of SHEN26 or its metabolites excreted in urine and feces (Ae).
fe After a Single Dose of SHEN26 capsule | From predose to 72 hours postdose
  (For SAD 400mg dose group only) The cumulative fraction of SHEN26 excreted in urine and feces (fe).
Cmax,ss After Multiple Doses of SHEN26 capsule | From predose to 48 hours postdose
  The maximum concentration at steady state (Cmax,ss) of SHEN26 capsule.
Cmin,ss After Multiple Doses of SHEN26 capsule | From predose to 48 hours postdose
  The minimum concentration at steady state (Cmin,ss) of SHEN26 capsule.
Cavg After Multiple Doses of SHEN26 capsule | From predose to 48 hours postdose
  The average concentration at steady state (Cavg) of SHEN26 capsule.
Tmax,ss After Multiple Doses of SHEN26 capsule | From predose to 48 hours postdose
  The time to the maximum concentration at steady state (Tmax,ss) of SHEN26 capsule.
AUCτ After Multiple Doses of SHEN26 capsule | From predose to 48 hours postdose
  The area under the concentration-time curve during the dosing interval (AUCτ) of SHEN26 capsule.
CLss/F After Multiple Doses of SHEN26 capsule | From predose to 48 hours postdose
  The apparent clearance at steady state (CLss/F) of SHEN26 capsule.
Vss/F After Multiple Doses of SHEN26 capsule | From predose to 48 hours postdose
  The apparent volume of distribution at steady state (Vss/F) of SHEN26 capsule.
DF After Multiple Doses of SHEN26 capsule | From predose to 48 hours postdose
  The degree of fluctuation in the concentration during the dosing interval (DF) of SHEN26 capsule.
Rac,AUC After Multiple Doses of SHEN26 capsule | From predose to 48 hours postdose
  The accumulation ratio based on AUC (Rac,AUC) of SHEN26 capsule.
Rac,Cmax After Multiple Doses of SHEN26 capsule | From predose to 48 hours postdose
  The accumulation ratio based on Cmax (Rac,Cmax) of SHEN26 capsule.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhao, MMed, Principal Investigator — The Second Hospital of Anhui Medical University; Wei Hu, MD, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun C, Liu H, Ouyang Z, Ding J, Zhang Q, Ma H, Xu D, Zhang Q, Zhou R, Yang M, Hu W. Safety, tolerability, and pharmacokinetics of the novel RdRp inhibitor SHEN26 against SARS-CoV-2: a randomized, placebo-controlled, double-blind Phase I study in healthy subjects. Expert Opin Investig Drugs. 2024 May;33(5):533-542. doi: 10.1080/13543784.2024.2347302. Epub 2024 Apr 30. PMID 38662639
- [Derived] Zhou Q, Yang S, Cao L, Yang Y, Xu T, Chen Q, Lu H, Li Y, Guo D, Zhang X. Preclinical characterization and anti-SARS-CoV-2 efficacy of ATV014: an oral cyclohexanecarboxylate prodrug of 1'-CN-4-aza-7,9-dideazaadenosine C-nucleoside. Signal Transduct Target Ther. 2023 Jan 12;8(1):27. doi: 10.1038/s41392-023-01310-0. No abstract available. PMID 36635259